CLINICAL TRIAL: NCT06401421
Title: EXActDNA-003 / NSABP B-64: Breast Cancer Clinical Validation Study to Predict Recurrence of High-Risk Early Breast Cancer Treated With Neoadjuvant Therapy Using a Bespoke Circulating Tumor DNA Assay to Detect Molecular Residual Disease
Brief Title: EXActDNA-003 / NSABP B-64: Study of Molecular Residual Disease Detection in Breast Cancer (MRD)
Status: Recruiting | Type: Observational
Sponsor: Exact Sciences Corporation (Industry)
Collaborators: NSABP Foundation Inc (Network)
Responsible Party: Sponsor
Other Study IDs: 2023-05
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; ctDNA
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- Participants with High Risk Early Breast Cancer: Participants with High Risk Early Breast Cancer
  Interventions: Diagnostic Test: ctDNA MRD test

INTERVENTIONS:
Diagnostic Test: ctDNA MRD test — Blood and tissue samples will be collected for the ctDNA MRD test
  Other Names: Oncodetect™

SUMMARY:
The EXActDNA-003 study will prospectively enroll participants who are planning to undergo chemotherapy for high-risk, early breast cancer, who are willing to provide tissue and blood specimens for circulating tumor DNA (ctDNA) analysis.

Participants will be followed for up to 5.5 years.

ELIGIBILITY:
Inclusion Criteria:

1. The participant or a legally authorized representative must provide study-specific informed consent prior to study entry.
2. The participant must be ≥ 18 years of age.
3. ECOG performance status 0 or 1.
4. Histologically confirmed invasive carcinoma of the breast.
5. Planned neoadjuvant therapy which includes cytotoxic chemotherapy.
6. Tumor size ≥ 2.1 cm in greatest diameter.
7. Unifocal or multifocal cancer documented to be the same histologic clinical subtype.
8. Clinically node positive or if node negative, any one of the following:

   1. TNBC or HER2+ subtype
   2. HR+/HER2-negative with at least one of the following:

   i. High tumor grade (G3) ii. Ki67 index of 20% or higher iii. High genomic risk (Oncotype DX® (ODX) Breast Recurrence Score of > 25, MammaPrint® High, etc.)
9. Willing and able to comply with the study requirements, which includes the collection of a total of 34 cc (2.5 Tablespoons) of blood for each research blood draw.
10. Available residual tissue from diagnostic biopsy from the breast or an involved ipsilateral lymph node for submission to create a bespoke ctDNA assay.

Exclusion Criteria:

1. Definitive clinical or radiologic evidence of metastatic disease.
2. Initiated neoadjuvant therapy for current breast cancer diagnosis.
3. Synchronous diagnosis of another invasive cancer, other than this breast cancer, except for non-melanoma skin cancers.
4. Completed all therapy (including endocrine therapy) <5 years ago for any previous invasive solid organ malignancy (with exception of non-melanoma skin cancers) including prior breast cancer. Individuals with a prior history of noninvasive (in situ) carcinomas may participate if they have received definitive treatment.
5. Completed all therapy for any previous hematologic malignancy < 5 years ago.
6. Multicentric or contralateral invasive breast cancers.
7. Known pregnancy at time of enrollment.
8. Prior solid organ transplant.
9. Prior allogeneic hematopoietic stem cell transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 who will undergo neoadjuvant treatment for high-risk, early breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Core biopsy tissue evaluability rate | 3 years
Distant Recurrence Free Interval (dRFI) | 6 years

SECONDARY OUTCOMES:
Prevalence of tumor mutations and germline variants | 6 years
Sensitivity/Specificity | 6 years
Prevalence of test positivity | 6 years
Pathologic complete response (pCR) status | 6 years
Recurrence-free interval (RFI) | 6 years
Invasive breast cancer-free survival (IBCFS) | 6 years
Event-free survival (EFS) | 6 years
Overall survival (OS) | 6 years
Lead Time | 6 years

CONTACTS AND LOCATIONS:
Locations (58):
- United States (53):
  - Katmai Oncology Group - Anchorage, Anchorage, Alaska
  - Stanford Cancer Institute, Palo Alto, California
  - Harbor-UCLA Medical Center - Hematology / Oncology, Torrance, California
  - Kaiser Permanente Medical Center, Vallejo, California
  - UCHealth Cancer Care - Anschutz Medical Campus - University of Colorado Cancer Center, Aurora, Colorado
  - AdventHealth East Altamonte Oncology and Hematology, Altamonte Springs, Florida
  - Mount Sinai Medical - Comprehensive Cancer Center, Miami Beach, Florida
  - Baptist Cancer Care - Plantation, Plantation, Florida
  - St. Joseph's Women's Hospital, Tampa, Florida
  - Rush Cancer Center, Chicago, Illinois
  - Deaconess Chancellor Center for Oncology, Newburgh, Indiana
  - University of Kansas Cancer Center, Westwood, Kansas
  - St. Elizabeth Edgewood Hospital, Edgewood, Kentucky
  - Norton Cancer Institute - Downtown, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Weinberg Center at Mercy, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - MedStar Georgetown Cancer Institute, Baltimore, Maryland
  - The Center for Cancer and Blood Disorders - Bethesda, Bethesda, Maryland
  - James M Stockman Cancer Institute, Frederick, Maryland
  - Tate Cancer Center at UM Baltimore Washington, Glen Burnie, Maryland
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - Holy Cross Hospital - Silver Spring, Silver Spring, Maryland
  - University of Maryland St. Joseph Medical Center, Towson, Maryland
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Metro Minnesota Community Oncology Consortium (MMCORC), Saint Louis Park, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Stony Brook Medicine, Stony Brook, New York
  - Atrium Health Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Cancer Institute - Elizabeth, Charlotte, North Carolina
  - FirstHealth Outpatient Cancer Center, Pinehurst, North Carolina
  - UNC Cancer Care at Nash, Rocky Mount, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Aultman Timken Family Cancer Center, Canton, Ohio
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - Penn State Health Medical Group - Andrews Patel, Harrisburg, Pennsylvania
  - Penn State Cancer Institute, Hershey, Pennsylvania
  - UPMC Magee - Womens Hospital, Pittsburgh, Pennsylvania
  - Guthrie Sayre, Sayre, Pennsylvania
  - Women & Infants Hospital, Providence, Rhode Island
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Ballad Health Cancer Center, Kingsport, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Joe Arrington Cancer Research & Treatment Center, Lubbock, Texas
  - Alan B. Pearson Regional Cancer Center, Lynchburg, Virginia
  - Bon Secours Cancer Institute at St. Francis, Midlothian, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - WVU Cancer Institute, Morgantown, West Virginia
  - Aurora Cancer Care - Wauwatosa, Wauwatosa, Wisconsin
- Canada (5):
  - Maisonneuve-Rosemont Hospital (HMR), Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health - Glen Site, Montreal, Quebec
  - Hôpital du Saint-Sacrement, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications of the study will be shared after deidentification. This may include test, tables, figured, and appendices. The study protocol, statistical analysis plan (when applicable), informed consent form (when applicable). May not be reproduced nor disseminated outside of Exact Sciences without permission and the clinical study report (when applicable) will also be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available from 2 years and ending 4 years after publication
Access Criteria: Proposals for access to data should be directed to clinicaltrials@exactsciences.com. To gain access, data requestors will need to provide a methodologically sound proposal and sign a data access agreement. Researchers are required to obtain necessary Institutional Review Board (IRB)/Institutional Ethics Committee (IEC) approvals or waivers as applicable to conduct research.